CLINICAL TRIAL: NCT05158777
Title: A Randomized, Blind, Controlled Clinical Trial to Evaluate Safety and Immunogenicity of Live Attenuated Varicella Vaccine After a Two-dose Vaccination Course in Healthy Population Aged ≥13 Years Old
Brief Title: Safety and Immunogenicity of Live Attenuated Varicella Vaccine in Healthy Population Aged ≥13 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020LP00094-III
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group with the immunization course of 0,28 days or 0,56 days (Experimental): 1240 subjects (including 620 children aged 13-17 years and 620 adults aged 18 years and older) will receive two doses of experimental vaccine with the immunization course of 0,28 days or 0,56 days.
  Interventions: Biological: Live attenuated varicella vaccines manufactured by Shanghai Institute of Biological Products Co.,Ltd.
- Control Group (Active Comparator): 1240 subjects (including 620 children aged 13-17 years and 620 adults aged 18 years and older) will receive two doses of control vaccine with the immunization course of 0,28 days or 0,56 days.
  Interventions: Biological: Live attenuated varicella vaccines manufactured by Changchun BCHT Biotechnology Co.,Ltd

INTERVENTIONS:
Biological: Live attenuated varicella vaccines manufactured by Shanghai Institute of Biological Products Co.,Ltd. — live varicella-zoster virus in 0.5 mL of sucrose, sodium chloride, potassium chloride, sodium glutamate, phosphate and injection water per injection
  Arms: Experimental Group with the immunization course of 0,28 days or 0,56 days
Biological: Live attenuated varicella vaccines manufactured by Changchun BCHT Biotechnology Co.,Ltd — live varicella-zoster virus in 0.5 mL of mannitol, dextrose tincture, sucrose, trehalose, human serum albumin and injection water per injection
  Arms: Control Group

SUMMARY:
This is a randomized, blind, controlled clinical trial of live attenuated varicella vaccines manufactured by Shanghai Institute of Biological Products Co.,Ltd. The purpose of this study is to evaluate the immunogenicity and safety of a two doses vaccination of investigational vaccine with 0,28 day and 0,56 day immunization schedule in population aged ≥13 years old.

DETAILED DESCRIPTION:
This study is a randomized, blind, controlled phase III clinical trial in population aged ≥13 years old. The experimental vaccine will be manufactured by Shanghai Institute of Biological Products Co.,Ltd.. A total of 2480 subjects aged 13 years and older will be enrolled with 1240 subjects in 13~17 years old group and1240 subjects in 18 years and older group. 1240 subjects in each age group would be randomly divided into experimental group and control group according to 1:1 ratio, and subjects will receive two doses of vaccine with the immunization course of 0,28 days or 0,56 days. In addition, 400 subjects from experimental group (100 subjects per subgroup) would be selected to collect blood at 3 and 5 years after immunization to evaluate immune persistence of live attenuated varicella vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy population aged 13 years and above;
* Proven legal identity;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 13-17 years, both subjects and guardians need to sign the informed consent form).

Exclusion Criteria:

* Disease history or vaccine history of chickenpox or shingles;
* Have fever before vaccination, axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 6 months;
* History of severe allergy and asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioedema and abdominal pain;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension (adult field measurement: SBP ≥140mmHg or diastolic blood pressure ≥90mmHg) that could not be controlled by drugs, diabetes, liver and kidney diseases, malignant tumors, etc.;
* Family history of psychosis,severe neurological disease (epilepsy, convulsions or twitching) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia, functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 6 months;
* Participating in other drug/vaccine clinical trial;
* Receipt of attenuated live vaccines in the past 28 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2480 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate of HI antibody | Day 42 after the whole schedule
  The seroconversion rate of the antibody 42 days among all subjects after the second vaccination.
GMT of HI antibody | Day 42 after the whole schedule
  The GMT of the antibody 42 days among all subjects after the second vaccination.

SECONDARY OUTCOMES:
Seroprotection rate of HI antibody | Day 42 after the whole schedule
  The seroprotection rate of the antibody 42 days among all subjects after the second vaccination.
Incidence of adverse reactions within 30 minutes after each dose | Within 30 minutes after each dose
  Incidence of adverse reactions within 30 minutes after each dose vaccination with immunization course of 0,28 days and 0,56 days.
Incidence of adverse reactions within 0~28 days after each dose | Within 0~28 days after each dose
  Incidence of adverse reactions within 0~28 days after each dose vaccination with immunization course of 0,28 days and 0,56 days.
Incidence of serious adverse events | From vaccination to 6 months after the second vaccination
  Incidence of serious adverse events from vaccination to 6 months after the second vaccination with immunization course of 0,28 days and 0,56 days

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Henan Provincial Center for Disease Prevention and Control, Zhenzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No